CLINICAL TRIAL: NCT03827551
Title: Preliminary Study of the Quality of the Oral Flora in Parkinson's Patients
Acronym: PARKIDENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Capionis (Unknown); France Parkinson Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2018/44
Record Dates: First submitted 2019-01-25; First posted 2019-02-01 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Oral Health; Parkinson Disease
Keywords: Oral Health; Parkinson Disease; Tooth cavities; Saliva; Mucosa
MeSH Terms: conditions — Parkinson Disease; Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parkinson's Patients (Experimental)
  Interventions: Behavioral: Delivery of oral hygiene advices

INTERVENTIONS:
Behavioral: Delivery of oral hygiene advices — Patients will benefit from hygiene advice and maintenance of good oral health. No treatment will be administered as part of this study. Patients will continue their usual treatment according to the contraindications. Patients will benefit from salivary sampling and a collection of oral bacteria contained in the dental plaque using paper tips. These reviews will be conducted during the Inclusion Visit and the 6 month Follow-Up Visit.

SUMMARY:
This is a prospective interventional clinical study whose main objective is to determine the impact of oral hygiene guidance on the oral health status of patients with Parkinson disease

DETAILED DESCRIPTION:
Caries and periodontitis are infectious diseases that can eventually lead to the loss of the dental organ. The masticatory deficit engendered will have repercussions on the general state of the subject and on his quality of life (pains, difficulties of feeding which can cause nutritional deficiencies ...). The systematic review of the literature, despite low levels of evidence, shows that there is an influence of Parkinson's disease on oral health. Our goal is therefore to determine the impact of implementing appropriate oral hygiene measures on improving the quality of life of patients with Parkinson's disease.

This is a 40-patient, interventional, preliminary study that will rely on indicators of oral health status (DMF, Periodontal Index, presence of pathogenic bacteria), as well as a questionnaire measuring impact of oral conditions on patient well-being (OHIP-14). These data will be collected before and after the implementation of the hygiene measures, within a period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Patient with Parkinson disease
* Able to give written informed consent
* Affiliated to French health care system

Exclusion Criteria:

* Patient under tutorship and curatorship
* Pregnant women
* Patient wearing subtotal or total dental prosthesis
* Antibiotic treatment or antiseptic mouthwashes in the month prior to sampling
* Patient with less than 6 teeth distributed on maxilla and mandible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-04-06 (Actual)

PRIMARY OUTCOMES:
Decayed Missing Filled (DMF) index score | 6 months after inclusion
  Min value : 0 (good oral health), Max value : 32
Presence of cariogenic bacteria in saliva and dental film | 6 months after inclusion
  Streptococcus mutans and Lactobacillus
Presence of periodontopathogenic bacteria in saliva and dental film | 6 months after inclusion
  Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Tannerella forsythia, Treponema denticola, Prevotella intermedia, Fusobacterium nucleatum, Peptostreptococcus micros, Eikenella corrodens, Campylobacter rectus

SECONDARY OUTCOMES:
Decayed Missing Filled (DMF) index score | Inclusion visit (Day 0)
  Min value : 0 (good oral health), Max value : 32
Presence of cariogenic bacteria in saliva and dental film | Inclusion visit (Day 0)
  Streptococcus mutans and Lactobacillus
Presence of periodontopathogenic bacteria in saliva and dental film | Inclusion visit (Day 0)
  Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Tannerella forsythia, Treponema denticola, Prevotella intermedia, Fusobacterium nucleatum, Peptostreptococcus micros, Eikenella corrodens, Campylobacter rectus
Change of Oral Health Impact Profile-14 (OHIP-14) | Inclusion Visit (Day 0) and 6 month after
  Min value : 14, Max value : 70 (satisfactory oral health)
Change of Geriatric/General Oral Health Assessment Index (GOHAI) | Inclusion Visit (Day 0) and 6 month after
  Min value : 12, Max value : 60 (satisfactory oral health)
Saliva pH | Inclusion Visit (Day 0) and 6 month after
  Normal / Acid / Very acid
Quantification of saliva flow | Inclusion Visit (Day 0) and 6 month after
  Normal / Low
Change of Community Periodontal Index of Treatment Needs (CPITN) | Inclusion Visit (Day 0) and 6 month after
  CPI Min value : 0 (healthy periodontium), Max value : 4 ; TN Min value : 0 (No periodontal treatment needed), Max value : 3

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Donnet L, Claisse O, Samot J. Serotype and distribution of adhesion genes in Streptococcus mutans isolated from people with Parkinson's disease. Odontology. 2025 Oct;113(4):1520-1532. doi: 10.1007/s10266-025-01078-5. Epub 2025 Mar 6. PMID 40048130